CLINICAL TRIAL: NCT01495936
Title: The Influence Of Continuous Positive Airway Pressure and Positive End-Expiratory Pressure, With A Recruitment Maneuver, On Oxygenation During One Lung Ventilation Employing A Lung Protective Ventilation Strategy.
Brief Title: The Effect of Two Airway Interventions, During One Lung Ventilation, on Blood Oxygen Content
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HSREB 18480
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Thoracic, Diseases
Keywords: One Lung Ventilation (OLV); Continuous Positive Airway Pressure (CPAP); Positive End Expiratory Pressure (PEEP); Lung recruitment maneuver; Hypoxia
MeSH Terms: conditions — Thoracic Diseases; Hypoxia | interventions — Positive-Pressure Respiration; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Positive Airway Pressure (Active Comparator): After 20 minutes ventilation on one lung (during anesthesia) the patient will be randomly assigned to the study arm "Continuous Positive Airway Pressure (CPAP)". CPAP will be applied for 20 minutes to the non-ventilated lung at a pressure of 5cmH20 using the disposable Mallinckrodt Bronchocath CPAP system.
  Interventions: Procedure: Continuous Positive Airway Pressure
- RM + Positive End Expiratory Pressure (Active Comparator): After 20 minutes of ventilation on one lung (during anesthesia) the patient will be randomly assigned to the study arm "RM + Positive End Expiratory pressure" which is a Recruitment Maneuver (RM) followed by Positive End Expiratory Pressure (RM-PEEP) which will be applied to the ventilating lung at a pressure of 5cmH2O.
  Interventions: Procedure: RM + Positive End Expiratory Pressure

INTERVENTIONS:
Procedure: RM + Positive End Expiratory Pressure — A recruitment maneuver (RM) will be applied to the ventilated lung by performing a valsalva maneuver for 5 seconds (holding the inspiratory pressure at 25cmH2O). Immediately after the RM, Positive End Expiratory Pressure (PEEP) will be applied to the ventilated lung at a pressure of 5cmH2O for 20 minutes. Both the RM and PEEP will be performed using the operating room ventilator.
  Arms: RM + Positive End Expiratory Pressure
Procedure: Continuous Positive Airway Pressure — Continuous positive airway pressure, at a pressure of 5cmH2O will applied to the non-ventilated lung for 20 minutes by the Mallinckrodt Bronchocath Disposable CPAP system (a recognised anesthetic breathing system design for CPAP)
  Arms: Continuous Positive Airway Pressure

SUMMARY:
Patients requiring one lung ventilation (OLV) for open thoracic surgery will be ventilated (breathing performed by a breathing machine) during anesthesia using a lung protective ventilation strategy (small breath volumes at 6ml/kg). During thoracic surgery the anesthesiologist is able to ventilate only one lung by inserting a special breathing tube, allowing the surgeon to operate on the non ventilated (diseased) lung. In a randomized trial two interventions used to improve blood oxygen levels during one lung ventilation will be compared . The two interventions are:

1. Continuous Positive Airway Pressure (CPAP) applied to the non ventilated (non breathing) lung and
2. Positive End Expiratory Pressure following a lung Recruitment Maneuver (RM-PEEP) to the ventilated (breathing) lung.

CPAP is performed by applying a steady flow of oxygen to the non ventilated (non breathing) lung at a continuous gentle pressure of 5cmH20.

To perform a Recruitment Maneuver (RM) the anesthesiologist inflates the ventilated (breathing) lung with oxygen, holding the breath for 25 seconds so all the lung is opened up. Immediately after the recruitment maneuver PEEP will be applied. PEEP is an action which also helps keep the lung open, maintaining the benefits achieved by the RM. It is performed by adjusting settings on the ventilator (breathing machine). The ventilator creates and applies a gentle pressure (5cmH20) to the ventilating lung at the end of each breath.

The outcome measure will be the oxygen content in blood (PaO2), measured in mmHg, using blood sample analysis.

The null hypothesis is that compared to CPAP, RM-PEEP does not significantly increase the oxygen content of blood during OLV when using a lung protective ventilation strategy.

DETAILED DESCRIPTION:
Patients requiring one lung ventilation (OLV) for open thoracic surgery will be ventilated intra-operatively using a lung protective ventilation strategy (small tidal volumes {Vts} at 6ml/kg Ideal Body Weight {IBW}). In a randomized, crossover trial Continuous Positive Airway Pressure (CPAP) to the non ventilated lung or a Recruitment Maneuver (RM) followed by the application of Positive End Expiratory Pressure (PEEP) (acronym RM-PEEP) to the ventilated lung will be applied and blood oxygenation (PaO2) measured by arterial blood gas sampling to determine which intervention has the most beneficial effect on PaO2 (CPAP or RM-PEEP).

CPAP will be applied at a pressure of 5cmH2O by a CPAP breathing circuit (designed for the purpose and commonly used in anesthetic practice). The PEEP will be applied at a pressure of 5cmH20 by the operating room (OR) anesthetic machine. The RM will involve a valsalva maneuver, held for 5 seconds at a pressure of 25cmH20, again performed using the OR anesthetic machine.

Null hypothesis: Compared to CPAP, RM-PEEP does not significantly increase PaO2 or reduce the incidence of hypoxia (oxygen blood saturation less than or equal to 90%), when employing a lung protective ventilation strategy.

This study is based on our previous research (citation 12, Badner et al) in which we compared CPAP to PEEP alone (omitting the recruitment maneuver). Here it was noted that CPAP to the non ventilated lung improved oxygenation more than PEEP to the ventilated lung (even though PEEP is an easier modality to provide), when employing a lung protective ventilation strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Competent to give consent to enroll in study
3. Booked for scheduled open thoracotomy which involves wedge resection, lobectomy or pneumonectomy requiring OLV
4. American Society of Anesthesia physical status score (ASA) 1-4

Exclusion Criteria:

1. Unable to give consent
2. Pregnant women
3. Inability to insert an arterial line
4. Presence of other significant pulmonary impairment (PaO2 on room air <50mmHg, PaCO2 >50mmHg or known pulmonary hypertension (mean PAP>25mmHg)
5. Presence of significant cardiovascular disease
6. Altered liver function (Child Pugh scale ≥B)
7. Patients with bullous lung disease. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-10-17 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Partial pressure of oxygen in blood | Day 1
  Time 0 (the patient is anesthetized and being ventilated on two lungs, just prior to the commencement of one lung ventilation). Time 20 minutes (patient has been ventilated on one lung for 20 minutes and immediately prior to instituting one of the two intervention arms). Time 40 minutes (following a period of 20 minutes on one intervention arm [either CPAP or RM-PEEP]. The patient will then enter second intervention arm). Time 60 minutes ( 20 minutes after second intervention arm [either CPAP or RM-PEEP])

SECONDARY OUTCOMES:
Hypoxia | Day 1
  The incidence of hypoxia (oxygen saturation falling below 90%, measured by pulse oximetry) throughout the entire study period will be recorded and correlated with the study stage.
Hypoxia intervention techniques | Day 1
  The incidence of necessary hypoxia (oxygen saturation below 90%) intervention techniques (performed by the attending anesthesiologist) will be recorded once the patient has been commenced on one lung ventilation. The interventions recorded will be
  1. The need to revert back to two lung ventilation
  2. The need to clamp the operative pulmonary artery
  3. The need to add CPAP to the non ventilated lung despite being in the RM-PEEP arm of the study.
  4. The need to add a RM-PEEP to the ventilated lung despite being in the CPAP arm of the study

CONTACTS AND LOCATIONS:
Overall Officials: Neal Badner, MD FRCP (C), Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Victoria Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Karzai W, Schwarzkopf K. Hypoxemia during one-lung ventilation: prediction, prevention, and treatment. Anesthesiology. 2009 Jun;110(6):1402-11. doi: 10.1097/ALN.0b013e31819fb15d. PMID 19417615
- [Background] Licker M, Diaper J, Villiger Y, Spiliopoulos A, Licker V, Robert J, Tschopp JM. Impact of intraoperative lung-protective interventions in patients undergoing lung cancer surgery. Crit Care. 2009;13(2):R41. doi: 10.1186/cc7762. Epub 2009 Mar 24. PMID 19317902
- [Background] Schilling T, Kozian A, Huth C, Buhling F, Kretzschmar M, Welte T, Hachenberg T. The pulmonary immune effects of mechanical ventilation in patients undergoing thoracic surgery. Anesth Analg. 2005 Oct;101(4):957-965. doi: 10.1213/01.ane.0000172112.02902.77. PMID 16192502
- [Background] Fernandez-Perez ER, Keegan MT, Brown DR, Hubmayr RD, Gajic O. Intraoperative tidal volume as a risk factor for respiratory failure after pneumonectomy. Anesthesiology. 2006 Jul;105(1):14-8. doi: 10.1097/00000542-200607000-00007. PMID 16809989
- [Background] Licker M, de Perrot M, Spiliopoulos A, Robert J, Diaper J, Chevalley C, Tschopp JM. Risk factors for acute lung injury after thoracic surgery for lung cancer. Anesth Analg. 2003 Dec;97(6):1558-1565. doi: 10.1213/01.ANE.0000087799.85495.8A. PMID 14633519
- [Background] Schultz MJ, Haitsma JJ, Slutsky AS, Gajic O. What tidal volumes should be used in patients without acute lung injury? Anesthesiology. 2007 Jun;106(6):1226-31. doi: 10.1097/01.anes.0000267607.25011.e8. PMID 17525599
- [Background] Michelet P, D'Journo XB, Roch A, Doddoli C, Marin V, Papazian L, Decamps I, Bregeon F, Thomas P, Auffray JP. Protective ventilation influences systemic inflammation after esophagectomy: a randomized controlled study. Anesthesiology. 2006 Nov;105(5):911-9. doi: 10.1097/00000542-200611000-00011. PMID 17065884
- [Background] Tusman G, Bohm SH, Sipmann FS, Maisch S. Lung recruitment improves the efficiency of ventilation and gas exchange during one-lung ventilation anesthesia. Anesth Analg. 2004 Jun;98(6):1604-1609. doi: 10.1213/01.ANE.0000068484.67655.1A. PMID 15155312
- [Background] Fan E, Wilcox ME, Brower RG, Stewart TE, Mehta S, Lapinsky SE, Meade MO, Ferguson ND. Recruitment maneuvers for acute lung injury: a systematic review. Am J Respir Crit Care Med. 2008 Dec 1;178(11):1156-63. doi: 10.1164/rccm.200802-335OC. Epub 2008 Sep 5. PMID 18776154
- [Background] Hoftman N, Canales C, Leduc M, Mahajan A. Positive end expiratory pressure during one-lung ventilation: selecting ideal patients and ventilator settings with the aim of improving arterial oxygenation. Ann Card Anaesth. 2011 Sep-Dec;14(3):183-7. doi: 10.4103/0971-9784.83991. PMID 21860189
- [Background] Cohen E, Eisenkraft JB, Thys DM, Kirschner PA, Kaplan JA. Oxygenation and hemodynamic changes during one-lung ventilation: effects of CPAP10, PEEP10, and CPAP10/PEEP10. J Cardiothorac Anesth. 1988 Feb;2(1):34-40. doi: 10.1016/0888-6296(88)90145-7. PMID 2979130
- [Background] Badner NH, Goure C, Bennett KE, Nicolaou G. Role of continuous positive airway pressure to the non-ventilated lung during one-lung ventilation with low tidal volumes. HSR Proc Intensive Care Cardiovasc Anesth. 2011;3(3):189-94. PMID 23439803